CLINICAL TRIAL: NCT02985567
Title: An Observational Study of the Use of Chloral Hydrate for Ophthalmic Procedures in Children
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Principal Investigator, David S. Friedman, Professor, Johns Hopkins University
Other Study IDs: 00086598
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Intraocular Pressure; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intraocular pressure evaluation: Intraocular pressure evaluation using Icare tonometer 25 minutes after sedation, and then every 10 minutes until sedation is complete
  Interventions: Other: Intraocular pressure evaluation
- Safety of sedation: Documentation of:
  1. The need for repeat dosing of chloral hydrate.
  2. The level of alertness of the patient at the end of sedation and the total time between induction and readiness for discharge
  3. Interventions required for the patient including administration of oxygen, and need for intubation.

INTERVENTIONS:
Other: Intraocular pressure evaluation — Intraocular pressure checked with Icare rebound tonometer at 25 minutes after induction, followed by every 10 minutes until sedation was complete.
  Groups: Intraocular pressure evaluation

SUMMARY:
The study involves a prospective evaluation of chloral hydrate sedation for the measurement of intraocular pressure in children ages one month to five years of age.

DETAILED DESCRIPTION:
This study will be a prospective, non-randomized trial of children 1 month to 5 years of age who are determined to require a sedation procedure at the King Khaled Eye Specialist Hospital (KKESH). There will be two parts to the consent process. Oral consent will be administered to subjects who are not undergoing eye pressure evaluation. These children have chloral hydrate sedation for imaging or other eye evaluations. For these children, we will prospectively monitor the success rate of chloral hydrate sedation such that a complete ophthalmic or imaging evaluation could be performed and will determine the proportion of adverse events that occur due to sedation including vomiting, respiratory distress or depression, alterations in vital signs beyond reference ranges for normal sleeping children, hypoxia with oxygen saturation <90%, and unplanned hospital admission. No testing will be performed for study purposes on these individuals.

For children undergoing sedation who will have intraocular pressure measurements for clinical care purposes, we will perform additional eye pressure measurements as part of the research protocol. Written consent will be obtained to allow us to additionally measure their intraocular pressure as specified below.

After recruitment and completion of informed consent procedures by parents, subjects' medical and ocular history will be reviewed by a study ophthalmologist and one of two pediatricians overseeing sedation procedures. Patients unable to undergo intraocular pressure measurement due to infection or ocular surface disease and those in whom chloral hydrate sedation is medically contraindicated will be excluded. Age, gender, diagnosis, current medications and surgical history will be recorded from the clinical chart for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* ages 1 month to five years
* require sedation for ophthalmic care

Exclusion Criteria:

* weight <3 kg or >20 kg
* infection/ocular surface disease
* medical contraindication of chloral hydrate
* green or gray nasal discharge
* fever, productive cough, chest retractions, or other signs of respiratory infection
* oxygen saturation < 90%
* active infectious disease such as rubella or varicella
* rectal or tympanic temperature > 37.7 degrees, or oral or temporal artery temperature > 37.2 degrees
* history of current ongoing vomiting and diarrhea
* anemia (Hgb < 9.0mg),
* history of seizure in past 6 weeks

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 month to five years requiring sedation for ophthalmic care at King Khaled Eye Specialist Hospital (KKESH).
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2013-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in intraocular pressure during chloral hydrate sedation | 25 minutes after sedation to 125 minutes after sedation
  Unit- mmHg

SECONDARY OUTCOMES:
Chloral hydrate dose required for successful sedation | Adminstration to adequate sedation (up to 30 minutes)
  Unit- mg
Time to recovery | Sedation induction to 125 minutes after sedation
  Unit- minutes
Hear rate under sedation | Sedation induction to 125 minutes after sedation
  Unit- beats per minute
Blood pressure under sedation | Sedation induction to 125 minutes after sedation
  Unit- mmHg
Oxygen saturation under sedation | Sedation induction to 125 minutes after sedation
  Unit- %
Adverse events related to chloral hydrate sedation | Sedation induction to 125 minutes after sedation
  Unit- number of events (that occur from the following list) Vomiting, subclinical respiratory depression, recovery agitation, oxygen desaturation, airway obstruction, failed sedation, bradycardia, tachycardia, hypotension, hypertension, seizure, aspiration, apnea, arrhythmia, cardiac arrest Unit- number of events (that occur from the following list) Vomiting, subclinical respiratory depression, recovery agitation, oxygen desaturation, airway obstruction, failed sedation, bradycardia, tachycardia, hypotension, hypertension, seizure, aspiration, apnea, arrhythmia, cardiac arrest Unit- number of events (that occur from the following list) Vomiting, subclinical respiratory depression, recovery agitation, oxygen desaturation, airway obstruction, failed sedation, bradycardia, tachycardia, hypotension, hypertension, seizure, aspiration, apnea, arrhythmia, cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: David S Friedman, MD, MPH, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- King Khaled Eye Specialist Hospital (KKESH), Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vade A, Sukhani R, Dolenga M, Habisohn-Schuck C. Chloral hydrate sedation of children undergoing CT and MR imaging: safety as judged by American Academy of Pediatrics guidelines. AJR Am J Roentgenol. 1995 Oct;165(4):905-9. doi: 10.2214/ajr.165.4.7676990.
- [Background] Litman RS, Soin K, Salam A. Chloral hydrate sedation in term and preterm infants: an analysis of efficacy and complications. Anesth Analg. 2010 Mar 1;110(3):739-46. doi: 10.1213/ANE.0b013e3181ca12a8. Epub 2009 Dec 23. PMID 20032023